CLINICAL TRIAL: NCT00956787
Title: Phase 2 Study of AR-67 (DB-67) in Myelodysplastic Syndrome(MDS)
Brief Title: Study of AR-67 (DB-67) in Myelodysplastic Syndrome (MDS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arno Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR67-IIS201; MDACC PROTOCOL NO. 2008-0530; NCT00930540 (obsolete NCT alias)
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2009-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — 7-tert-butyldimethylsilyl-10-hydroxycamptothecin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with AR-67 (Experimental): Patients will receive AR-67 at an initial dose of 7.5 mg/m2 IV over 1 hour daily for 5 days.
  Interventions: Drug: AR-67 (20S)-7-t-Butyldimethylsilyl-10-hydroxycamptothecin)

INTERVENTIONS:
Drug: AR-67 (20S)-7-t-Butyldimethylsilyl-10-hydroxycamptothecin) — Patients will receive AR-67 at an initial dose of 7.5 mg/m2 IV over 1 hour daily for 5 days. In patients with stable disease, treatment may continue for up to a total of 12 courses of therapy; about 1 to 2 years.
  Other Names: AR-67; (20S)-7-t-Butyldimethylsilyl-10-hydroxycamptothecin)

SUMMARY:
The purpose of this study is to determine if AR-67 is effective in the treatment for patients with MDS.

DETAILED DESCRIPTION:
The management of MDS has been, until recently, based mostly on supportive care. This includes transfusion support, hematopoietic growth factors, and management of complications. With this management, the disease would run its natural course and the patient eventually died either from progression to acute leukemia or from complications associated with MDS itself (e.g., infections, hemorrhage). Recently, hypomethylating agents have offered promise for the management of patients with MDS. Although both agents have shown efficacy in a subset of patients, responses are usually either partial or hematologic improvement only, with CR rates <10%. In addition, responses have a median duration of less than 12 months. Thus, although both of these agents have improved the outcome of patients with MDS and been approved by the FDA for this purpose, there is clearly need for additional and more effective agents for this disease.

In vitro data suggested that topoisomerase I inhibitors could have activity in MDS, and a prolonged exposure appeared to be particularly effective. Topotecan was the first agent of this class explored for this purpose. A phase I study established the maximum tolerated dose (MTD) at 2 mg/m2/day as a continuous infusion for 5 days. Using this dose, a phase II study in patients with MDS and CMML, a complete remission rate of 31% was achieved. These agents are now considered the most effective available to date in the treatment of MDS and constitute standard therapy. Because of the different times when the studies were conducted and the different eligibility criteria used (e.g., patients with secondary MDS not eligible for decitabine, only patients with high-risk MDS eligible for topotecan), comparisons are somehow limited. However, results with topotecan compare favorably to those obtained with both 5-azacytidine and decitabine. The CR rate is the highest achieved with any of these agents. Response duration is shorter than that reported for AZA, but the remission duration for AZA includes hematologic improvements which constitute most of the responses with AZA. In addition, the AZA study continued therapy until the response was lost, while the topotecan study (as well as the decitabine study) administered by design only 4-6 cycles of therapy. Survival was shorter for patients treated with topotecan, but this is not unexpected considering that this population included 50% of patients with CMML and 32% with secondary MDS, both important adverse prognostic characteristics in MDS. The AZA study had the best survival, but it included 37% patients with RA or RAES and only 20% with intermediate-2 or high IPSS. Because the eligibility included patients with greater than 10% blasts, all MDS patients would have had a score of at least 1.5 and thus be classified in the intermediate-2 risk group.

Based on the favorable activity of topotecan as a single agent, topotecan was also used in combination with cytarabine in high-risk MDS (i.e., RAEB with >10% blasts or RAEBt). A CR rate of 56% was achieved, with a low rate of induction mortality (7%) in a population with a median age of 68 years. These results were at least equivalent to those achieved with an idarubicin and cytarabine combination both in a retrospective comparison of two different trials, and in a prospective randomized trial.

Overall, these results suggest that additional exploration of topoisomerase I inhibitors in myelodysplastic syndrome is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either of the following diagnoses:

   * MDS and >5% blasts, or IPSS risk group intermediate-1, intermediate-2 or high risk
   * Chronic myelomonocytic leukemia (CMML)
2. Patients must have failed prior therapy with either a hypomethylating agent (e.g., azacytidine, decitabine) alone or in combination with other agents. Patients with abnormalities in chromosome 5q, should have failed either a hypomethylating agent or lenalidomide.

   * Patients intolerant or unable to receive these agents will be considered eligible.
3. Age > 18 years. Because no dosing or adverse event data are currently available on the use of AR-67 in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
4. ECOG performance status 0-2.
5. Patients must have normal organ function as defined below:

   * Total bilirubin: < 1.5 x institutional upper limit of normal
   * ALT (SGPT): < 2.5 X institutional upper limit of normal
   * Creatinine: < 1.5 x institutional upper limit of normal
6. The effects of AR-67 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential (i.e., not post-menopausal for at least 12 months and not surgically sterile) and men must agree to use effective methods of contraception. Women of childbearing potential (any women who is not surgically sterile or > 2 years post menopause) must give consent for using a reliable method of contraception (e.g. double-barrier, tubal ligation or stable hormonal contraception) throughout the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Patients must have been off chemotherapy for 2 weeks prior to entering this study unless there is evidence of rapidly progressive disease. Patients must have recovered from the toxic effects of prior therapy to grade ≤1. The use of hydroxyurea is allowed to control counts up to 24 hrs prior to the start of therapy with AR-67.

Exclusion Criteria:

1. Nursing or pregnant females or females who plan pregnancy during the duration of the study.
2. Active and uncontrolled systemic infections.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the efficacy of AR-67 in treating patients with MDS who have failed prior therapies | 4 cycles (approximately 16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States